CLINICAL TRIAL: NCT03266809
Title: Longitudinal Characterisation of Cardiac Function in Recently-diagnosed Breast Cancer Patients
Brief Title: CARdiac Function Evaluation in Breast Cancer Patients
Acronym: CARE-B
Status: Completed | Type: Observational
Sponsor: Swansea University (Other)
Collaborators: Abertawe Bro Morgannwg University Health Board (Other)
Responsible Party: Principal Investigator, Prof Michael Lewis, Professor, Swansea University
Other Study IDs: 188676
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer Female
Keywords: Cardiac function; Cardio-toxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer Patients: Eligible participants will be women aged 18 years or over who have the following main characteristics:
  * Early invasive breast cancer (stage I-III)
  * Due to start SAT (adjuvant or neoadjuvant chemotherapy +/- trastuzumab +/- pertuzumab)
  * WHO performance status 0-2.

SUMMARY:
This study will investigate the influence of systemic adjuvant/neoadjuvant therapy (SAT: chemotherapy +/- anti-HER2 antibodies (trastuzumab +/- pertuzumab) on heart function/rhythm and cardio-respiratory fitness in recently diagnosed breast cancer patients. In some patients, SAT damages the heart (so-called 'cardiotoxicity') and this can have a serious impact on the patient's quality of life and overall survival. It has also been suggested that anticancer therapies may lead to repolarization abnormalities, QT prolongation and autonomic dysfunction, clinically reflected by an increase in HR and a reduction in heart rate variability (HRV). There is a lack of information in the literature regarding the extent and time-course of changes in cardiac function, cardiac rhythm and cardio-respiratory performance ('fitness') in these patients. Moreover, the differential influences of specific treatment regimes (e.g. SAT or SAT plus radiotherapy) and different chemotherapy drugs on cardio-respiratory performance remain unclear. A better understanding of these issues is the primary aim of this study.

DETAILED DESCRIPTION:
This study will focus on the following:

1. Cardiac function assessment: The conventional method for assessing heart function (in terms of 'ejection fraction') in patients being treated for cancer uses nuclear medicine (MUGA scan). MRI can also provide this information but it is not typically used for cardiac function assessment in these patients. MUGA scans are typically performed before chemotherapy in selected patients at higher risk of cardiotoxicity and in all cases before starting anti-HER2 antibody treatment (trastuzumab, pertuzumab). Patients receiving anti-HER2 antibody treatment receive repeat cardiac assessments at 3-4 month intervals until the completion of treatment - it is not practical or cost-effective to scan more frequently. This study will determine whether an alternative and inexpensive method for monitoring heart function (Impedance Cardiography, ICG) can adequately quantify changes in ejection fraction during treatment. If it can, then this technique could be used more frequently during and following treatment, with the aim of determining the treatment stages during which the heart is most at risk of damage. The ability of ICG to dynamically characterise a relatively rapid decline in cardiac function in breast cancer patients has not been established. Neither has its performance been compared with MRI or MUGA in this population. This study will investigate whether ICG is a sufficiently accurate and reliable alternative to MRI/MUGA for determining cardiac dysfunction during and following cancer treatment.
2. Cardiac rhythm and autonomic function assessment: Heart rate variability (HRV) reflects the modulation of the heart by the autonomic nervous system, and it can be quantified using several different methods based on analysis of the temporal changes between successive heartbeats. The development of autonomic dysfunction in breast cancer patients has been shown in a few small clinical studies, but the majority of these studies have considered HR rather than HRV, which is a much less robust measure of autonomic function. The few studies that have used HRV analysis have demonstrated significant reductions in HRV following the completion of anthracycline-based therapy. Previous research on other ECG markers (e.g. QT and QRS duration) in breast cancer patients has mainly focused on anthracycline-based regimes; the influence of trastuzumab treatment on ECG makers has been evaluated in only two studies to date. It is still not clear whether these changes can predict subsequent LV dysfunction although QT variability is a possible marker of myocardial contractility and has been shown to increase as a result of anthracycline therapy in breast cancer patients. This study aims to characterise the impact of different treatment regimes on the temporal properties of the ECG and will compare beat-to-beat QT variability and beat-to-beat T wave variability in breast cancer patients receiving a range of treatment regimes.
3. Body composition and cardiorespiratory fitness assessment: This study also aims to characterise the patterns of change in body composition, physical activity and cardiorespiratory fitness in breast cancer patients. The study will examine whether these modifiable factors might influence a patient's susceptibility to cardiac changes during treatment and, in turn, how these factors are affected by treatment. Of particular interest, it has been suggested that cardiorespiratory fitness (measured by the rate of oxygen uptake) is impaired in breast cancer patients compared to healthy controls, even seven years following the completion of treatment. Oxygen-uptake analysis will be performed in this study to explore possible compensatory mechanisms for abnormal pathology- or treatment-induced cardiac function in breast cancer patients. Fitness, physical activity and body composition will be assessed quantitatively using a range of objective techniques, including cardiopulmonary exercise testing on a cycle ergometer (fitness) with breath-by-breath gas analysis (cardiorespiratory function), accelerometery (activity levels) and DEXA radiography scans (body composition).

The main research questions in this study are:

1. Is the CARE-B protocol practically feasible and tolerable to early-stage breast cancer patients?
2. What is the level of agreement between cardiac (ventricular) function determined using cardiac MRI, MUGA and Impedance Cardiography in breast cancer patients receiving SAT?
3. Is cardiac rhythm (heart rate and QT variability) altered in breast cancer patients receiving SAT?
4. Is oxygen transport and oxygen uptake into tissue altered in breast cancer patients receiving SAT?
5. Does a patient's baseline physical activity, fitness and body composition affect their susceptibilities to treatment-induced cardio-respiratory problems?
6. Does a patient's physical activity, physical fitness and body composition change appreciably during SAT in these patients?

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be women aged 18 years or over with the following characteristics:

* Early invasive breast cancer (stage I-III)
* Due to start adjuvant or neoadjuvant therapy including either anthracycline-based chemotherapy, or chemotherapy + trastuzumab +/- pertuzumab
* WHO performance status <=2
* Absence of major cardiovascular or chronic respiratory problems, or other conditions that in the opinion of the clinician would contraindicate the use of physical exercise assessments
* Absence of contraindications for MRI scans, as listed in Paragraph 3.3. Patients unsuitable or unwilling to undergo MRI scans will be eligible for the study only if they are planned to receive trastuzumab, since this will include LVEF monitoring with MUGA scans or echocardiograms as part of routine care
* Provision of signed informed consent.

Exclusion Criteria:

* Presence of major cardiovascular or chronic respiratory problems, or other conditions that in the opinion of the clinician would contraindicate the use of treadmill exercise assessments
* Presence of contraindications for MRI scans:

  * Internal electronic devices such as neurostimulators or defibrillators
  * Replacement heart valve
  * Cardiac pacemaker
  * Intracranial vessel clips
  * Internal ear implant
  * Claustrophobia
  * Pregnancy.

MRI scans will be requested by a clinician after the exclusion of the above contraindications. Patients unsuitable or unwilling to undergo MRI scans will be eligible for the study only if they are planned to receive trastuzumab, since this includes LVEF monitoring with MUGA scans or echocardiograms as part of routine care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women aged 18 years or older who have early invasive breast cancer and who are due to begin adjuvant or neoadjuvant therapy for this condition, but who are otherwise free of major cardiovascular or chronic respiratory disease and who are capable of undertaking physical exercise.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Cardiac Function (stroke volume or ejection fraction) | At completion of treatment, an average of 13 months
  Cardiac function during/following treatment in breast cancer patients.
Cardiac Rhythm (heart rate variability) | At completion of treatment, an average of 13 months
  Cardiac rhythm during/following treatment in breast cancer patients.

SECONDARY OUTCOMES:
Physical activity level (accelerometer-based activity level 'counts') | At completion of treatment, an average of 13 months
  Physical activity level during/following treatment in breast cancer patients.
Cardiorespiratory function (rate of respiratory oxygen uptake) | At completion of treatment, an average of 13 months
  Cardiorespiratory function during/following treatment in breast cancer patients.
Body mass composition (from DEXA scan) | At completion of treatment, an average of 13 months
  Body fat mass and fat-free mass, and bone mineral density

CONTACTS AND LOCATIONS:
Overall Officials: Professor Lewis, Study Director — Swansea University
Locations (1):
- Singleton Hospital, Swansea, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No